CLINICAL TRIAL: NCT02209532
Title: A Randomized, Prospective, Open Label, Multicenter Study Assessing the Safety and Utility of PINPOINT® Near Infrared Fluorescence Imaging in the Identification of Lymph Nodes in Patients With Uterine and Cervical Malignancies Who Are Undergoing Lymph Node Mapping
Brief Title: A Study Assessing the Safety and Utility of PINPOINT® Near Infrared Fluorescence Imaging in the Identification of Lymph Nodes in Patients With Uterine and Cervical Malignancies Who Are Undergoing Lymph Node Mapping
Acronym: FILM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novadaq Technologies ULC, now a part of Stryker (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PP LNM 01
Record Dates: First submitted 2014-07-29; First posted 2014-08-06 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Endometrial Cancer; Uterine Cancer; Cervical Cancer
Keywords: Lymph node mapping; Endometrial cancer; Uterine cancer; Cervical cancer
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blue - PINPOINT (Active Comparator): The cervix will be injected 4 times with a 1ml solution of 1% Isosulfan blue followed by injection 4 times of 1 ml of 1.25 mg/ml solution of ICG. LN mapping with Blue dye will be performed until the investigator identifies all blue nodes or determines that blue nodes cannot be identified. Once complete, the Investigator will begin mapping with PINPOINT until all 'ICG' nodes are identified or the investigator determines that 'ICG' nodes cannot be identified. Once mapping with both Blue dye and PINPOINT have been completed and documented, LNs identified with Blue dye or PINPOINT will be excised.
  Interventions: Device: PINPOINT
- PINPOINT - Blue (Active Comparator): The cervix will be injected 4 times with 1 ml of a 1.25 mg/ml solution of ICG followed by injection 4 times of a 1 ml solution of 1% Isosulfan blue. LN mapping with PINPOINT will be performed until the investigator identifies all 'ICG' nodes or determines that 'ICG' nodes cannot be identified. Once complete, the Investigator will begin mapping with Blue dye until all 'blue' nodes are identified or the investigator determines that 'blue' nodes cannot be identified. Once mapping with both Blue dye and PINPOINT have been completed and documented, LNs identified with Blue dye or PINPOINT will be excised.
  Interventions: Device: PINPOINT

INTERVENTIONS:
Device: PINPOINT — PINPOINT® Near Infrared Fluorescence Imaging to identify lymph nodes

SUMMARY:
This is a randomized, prospective, open label, multicenter study to assess the safety and utility of PINPOINT® Near Infrared Fluorescence Imaging (PINPOINT) in identification of lymph nodes (LN) in patients with uterine and cervical malignancies who are undergoing LN mapping.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Subjects with FIGO Clinical Stage I endometrial cancer undergoing minimally invasive hysterectomy with lymph node mapping.
* Subjects with FIGO Clinical Stage IA cervical cancer ≤ 2 cm in size undergoing minimally invasive hysterectomy, trachelectomy, or conization with lymph node mapping. Subjects with clinical Stage IA1 cervical cancer without lympho vascular space involvement (LVSI) and negative margins on cone biopsy are not to be included.
* Subjects with negative nodal status (N0)
* Subjects with negative metastatic involvement (M0).

Exclusion Criteria:

* Have had prior dissection and/or radiation in pelvis.
* Advanced cervical or endometrial cancer, T3/T4 lesions
* Diagnosis of cervical cancer with a tumor size greater than 2 cm.
* Locally advanced or inflammatory cervical or uterine cancer
* Metastatic cervical or uterine cancer.
* Known allergy or history of adverse reaction to ICG, iodine or iodine dyes.
* Known allergy or history of adverse reaction to Blue dye (Isosulfan blue) or triphenylmethane.
* Hepatic dysfunction defined as MELD Score > 12.
* Renal dysfunction defined as serum creatinine ≥ 2.0 mg/dl.
* Subjects who have participated in another investigational study within 30 days prior to surgery.
* Pregnant or lactating subjects.
* Subjects who, in the Investigator's opinion, have any medical condition that makes the subject a poor candidate for the investigational procedure, or interferes with the interpretation of study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frumovitz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (8):
- United States (5):
  - O'Connor Hospital, San Jose, California
  - Lee Memorial Hospital, Fort Myers, Florida
  - Memorial Sloan Kettering, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - CHU de Québec - Université Laval, Québec, Quebec
- Hospital HIMA San Pablo, Caguas, Puerto Rico

REFERENCES:
- [Derived] Frumovitz M, Plante M, Lee PS, Sandadi S, Lilja JF, Escobar PF, Gien LT, Urbauer DL, Abu-Rustum NR. Near-infrared fluorescence for detection of sentinel lymph nodes in women with cervical and uterine cancers (FILM): a randomised, phase 3, multicentre, non-inferiority trial. Lancet Oncol. 2018 Oct;19(10):1394-1403. doi: 10.1016/S1470-2045(18)30448-0. Epub 2018 Aug 22. PMID 30143441

RESULTS

PARTICIPANT FLOW:
Groups:
- Lymph Node Mapping With Isosulfan Blue Followed by PINPOINT: The cervix will be injected 4 times with a 1ml solution of 1% Isosulfan blue followed by injection 4 times of 1 ml of 1.25 mg/ml solution of ICG. LN mapping with Blue dye will be performed until the investigator identifies all blue nodes or determines that blue nodes cannot be identified. Once complete, the Investigator will begin mapping with PINPOINT until all 'ICG' nodes are identified or the investigator determines that 'ICG' nodes cannot be identified. Once mapping with both Blue dye and PINPOINT have been completed and documented, LNs identified with Blue dye or PINPOINT will be excised.
  PINPOINT: PINPOINT® Near Infrared Fluorescence Imaging to identify lymph nodes
- Lymph Node Mapping With PINPOINT Followed by Isosulfan Blue: The cervix will be injected 4 times with 1 ml of a 1.25 mg/ml solution of ICG followed by injection 4 times of a 1 ml solution of 1% Isosulfan blue. LN mapping with PINPOINT will be performed until the investigator identifies all 'ICG' nodes or determines that 'ICG' nodes cannot be identified. Once complete, the Investigator will begin mapping with Blue dye until all 'blue' nodes are identified or the investigator determines that 'blue' nodes cannot be identified. Once mapping with both Blue dye and PINPOINT have been completed and documented, LNs identified with Blue dye or PINPOINT will be excised.
  PINPOINT: PINPOINT® Near Infrared Fluorescence Imaging to identify lymph nodes
Period: Overall Study
Arm/Group | Lymph Node Mapping With Isosulfan Blue Followed by PINPOINT | Lymph Node Mapping With PINPOINT Followed by Isosulfan Blue
Started | 90 | 90
Completed | 87 | 89
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: 180 subjects were randomized. 4 subjects were found to be ineligible after randomization (subjects did not receive study treatment) therefore, 176 subjects were included in the Baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Blue - PINPOINT | PINPOINT - Blue | Total
Number analyzed (Participants) | 87 | 89 | 176
Age, Customized [Count of Participants; unit: Participants]
  30-39 | 3 | 4 | 7
  40-49 | 6 | 4 | 10
  50-59 | 20 | 26 | 46
  60-69 | 33 | 41 | 74
  70-79 | 20 | 12 | 32
  >80 | 5 | 2 | 7
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 87 | 89 | 176
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 66 | 73 | 139
  Black or African American | 5 | 2 | 7
  Asian | 4 | 2 | 6
  Other | 2 | 0 | 2
Smoking Status [Count of Participants; unit: Participants]
  Never | 66 | 65 | 131
  Current | 2 | 5 | 7
  Past | 19 | 19 | 38
Alcohol Consumption [Count of Participants; unit: Participants]
  Yes | 34 | 31 | 65
  No | 53 | 58 | 111
ASA Classification [Count of Participants; unit: Participants]
  I - A normal healthy patient | 10 | 11 | 21
  II - A patient with mild systemic disease | 38 | 39 | 77
  III - A patient with severe systemic disease | 34 | 32 | 66
  Unknown ASA Classification | 5 | 7 | 12
Preoperative Diagnosis [Count of Participants; unit: Participants]
  Stage 1 Endometrial Cancer | 84 | 85 | 169
  Stage 1 Cervical Cancer | 2 | 2 | 4
  Stage 1A Cervical Cancer | 3 | 2 | 5
Endometrial Cancer Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 71 | 75 | 146
  Serous Carcinoma | 7 | 6 | 13
  Clear Cell Carcinoma | 4 | 0 | 4
  Carcinosarcoma | 1 | 2 | 3
  Other | 1 | 2 | 3
Cervical Cancer Histology [Count of Participants; unit: Participants]
  Squamous Cell Carcinoma | 0 | 3 | 3
  Adenocarcinoma | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of PINPOINT and IC2000 in the Identification of Lymph Nodes Defined as the Proportion of Confirmed Lymph Nodes Identified
Description: To assess the effectiveness of intraoperative PINPOINT Near Infrared Fluorescence Imaging in the identification of lymph nodes in subjects with uterine and cervical malignancies who are undergoing lymph node mapping.
Time Frame: Day 0
Population: All analyses were completed using the number of lymph nodes identified.
Measure: Number; unit: Confirmed Lymph Nodes
Units Other Than Participants: Confirmed Lymph Nodes
Arm/Group | PINPOINT - Blue | Blue - PINPOINT
Number analyzed (Participants) | 82 | 81
Number analyzed (Confirmed Lymph Nodes) | 238 | 247
Confirmed Lymph Nodes | 232 | 239

2. Secondary Outcome: Effectiveness of PINPOINT and Blue Dye in the Identification of at Least One Lymph Node Defined as the Number of Subjects in Which at Least One Confirmed Lymph Node Was Identified With Either PINPOINT or Blue Dye
Description: To evaluate the effectiveness of PINPOINT and Blue dye in the identification of at least one lymph node (confirmed to be lymphoid tissue) per subject.
Time Frame: Day 0
Population: 180 subjects were randomized. 4 subjects were found to be ineligible after randomization (subjects did not receive study treatment). Of the 176 subjects randomized who completed the study, 13 had significant protocol deviations. Thus, 163 subjects are included in the analysis population (81 subjects in the B-P arm and 82 subjects in the P-B arm).
Measure: Number; unit: Number of Subjects
Groups:
- PINPOINT-Blue: The cervix will be injected 4 times with 1 ml of a 1.25 mg/ml solution of ICG followed by injection 4 times of a 1 ml solution of 1% Isosulfan blue. LN mapping with PINPOINT will be performed until the investigator identifies all 'ICG' nodes or determines that 'ICG' nodes cannot be identified. Once complete, the Investigator will begin mapping with Blue dye until all 'blue' nodes are identified or the investigator determines that 'blue' nodes cannot be identified. Once mapping with both Blue dye and PINPOINT have been completed and documented, LNs identified with Blue dye or PINPOINT will be excised.
  PINPOINT: PINPOINT® Near Infrared Fluorescence Imaging to identify lymph nodes
Arm/Group | PINPOINT-Blue | Blue - PINPOINT
Number analyzed (Participants) | 82 | 81
Number of Subjects
  IC2000 and PINPOINT | 80 | 79
  Isosulfan Blue | 64 | 60

3. Secondary Outcome: Effectiveness of PINPOINT and Blue Dye in the Identification of Bilateral Lymph Nodes Defined as the Number of Subjects in Which Lymph Nodes Were Identified Bilaterally With Either PINPOINT or Blue Dye.
Description: To evaluate the effectiveness of PINPOINT and Blue dye in the identification of bilateral lymph nodes (confirmed to be lymphoid tissue).
Time Frame: Day 0
Population: as for outcome 2
Measure: Number; unit: Number of Subjects
Arm/Group | PINPOINT-Blue | Blue - PINPOINT
Number analyzed (Participants) | 82 | 81
Number of Subjects
  IC2000 and PINPOINT | 64 | 60
  Isosulfan Blue | 24 | 25

4. Secondary Outcome: Identification of Lymph Nodes Following Lymphatic Channels Defined as the Number of Subjects in Which Confirmed Lymph Nodes Were Identified by Following a Lymphatic Channel With Either PINPOINT or Blue Dye.
Description: To determine the proportion of lymph nodes identified from following lymphatic channels
Time Frame: Day 0
Population: as for outcome 2
Measure: Number; unit: Number of Subjects
Arm/Group | PINPOINT-Blue | Blue - PINPOINT
Number analyzed (Participants) | 82 | 81
Number of Subjects
  IC2000 and PINPOINT | 6 | 3
  Isosulfan Blue | 8 | 6

5. Secondary Outcome: Safety of Interstitial Injection of ICG Defined as the Number of Adverse Effects Related to ICG
Description: To assess the safety of interstitial injection of ICG for intraoperative lymphatic mapping, as measured by number of subjects experiencing adverse effects related to the study treatment.
Time Frame: Day 0 to Day 30
Population: as for outcome 2
Measure: Number; unit: Number of subjects
Arm/Group | PINPOINT-Blue | Blue - PINPOINT
Number analyzed (Participants) | 89 | 87
Number of subjects | 0 | 0

6. Secondary Outcome: Anatomic Distribution of Lymph Nodes
Description: To determine the anatomic distribution of lymph nodes
Time Frame: Day 0
Population: as for outcome 2
Measure: Number; unit: confirmed lymph nodes
Units Other Than Participants: Lymph Nodes
Arm/Group | PINPOINT-Blue | Blue - PINPOINT
Number analyzed (Participants) | 82 | 81
Number analyzed (Lymph Nodes) | 232 | 239
confirmed lymph nodes
  Left obturator/internal iliac | 28 | 36
  Left external iliac | 69 | 67
  Left common iliac | 11 | 6
  Right obturator/internal iliac | 39 | 45
  Right external iliac | 52 | 50
  Right common iliac | 17 | 18
  Presacral | 2 | 5
  Para-aortic node below IMA | 4 | 5
  Other | 10 | 7

ADVERSE EVENTS:
Time Frame: 30 Days
Description: Adverse Events were not monitored/assessed for each intervention separately. Both interventions (ICG/PINPOINT and Isosulfan Blue) were administered at the time of the adverse events.
Arm/Group | Blue - PINPOINT | PINPOINT - Blue
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/89
Serious Adverse Events (participants affected / at risk) | 4/87 | 1/89
Other Adverse Events (participants affected / at risk) | 13/87 | 10/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blue - PINPOINT (N=87) | PINPOINT - Blue (N=89)
Partial bowel obstruction (Gastrointestinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Trace pleural effusions (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blue - PINPOINT (N=87) | PINPOINT - Blue (N=89)
Procedural Pain (Injury, poisoning and procedural complications) | 13 | 10
Nausea (Gastrointestinal disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT02209532/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT02209532/SAP_001.pdf